CLINICAL TRIAL: NCT01514708
Title: The Safety and Immune Response to Influenza Vaccination in Pregnant Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Adimmune Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FLU11T12P
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2012-12

CONDITIONS: Influenza
Keywords: Influenza; Vaccination; Vaccine; Pregnancy
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AdimFlu-S Influenza Vaccine, 0.5mL/dose, receive 1 dose (Experimental)
  Interventions: Biological: AdimFlu-S Influenza Vaccine

INTERVENTIONS:
Biological: AdimFlu-S Influenza Vaccine — Suspension for injection

SUMMARY:
The purpose of this study is to evaluate the antibody response to the influenza vaccine (AdimFlu-S), as measured by hemagglutination inhibition (HAI) at 4 weeks post immunization in pregnant women in compliance with the requirements of the current European Union (EU) recommendations for the evaluation of the immunogenicity for a new formulation of a licensed flu vaccine (CPMP/BWP/214/96). Besides, the vaccine safety will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant female aged ≥ 18 years old.
2. Subject is pregnant for at least 3 months, inclusive.
3. Subject is willing and able to adhere to visit schedules and all study requirements.
4. Subject has read and signed the study-specific informed consent.

Exclusion Criteria:

1. Subject with previous complicated pregnancy or preterm delivery, spontaneous or medical abortion;
2. Subject with history or concurrent high risk of dangerous gestation such as gestational diabetes mellitus (GDM), pregnant induced hypertension, or preeclampsia;
3. Subject received any influenza vaccine within the previous 6 months;
4. Subject has a history of hypersensitivity to eggs or egg protein or similar pharmacological effects to study vaccine;
5. Subject or her family has the history of Guillain-Barré Syndrome;
6. Subject has current upper respiratory illness (URI), including the common cold or nasal congestion within 72 hours;
7. Subject with influenza-like illness as defined by the presence of fever (temperature over 38ºC) and at least two of the following four symptoms: headache, muscle/joint aches and pains (e.g. myalgia/arthralgia), sore throat and cough;
8. Subject receive any treatment with an investigational drug or device, or participation in a clinical study, within 3 months before consent;
9. Subject has immunodeficiency or is under immunosuppressive treatment.
10. Subject received any vaccine within 1 week prior to study vaccination or expected to receive one within 1 week after study vaccination;
11. Subject received any blood products, including immunoglobulin, in the past 3 months before consent;
12. Subject has underlying condition in the investigators' opinion may interfere with evaluation of the vaccine;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the seroprotection rate which is defined as the proportion of subjects with HAI titer ≥ 1:40. The other immunogenicity endpoints include seroconversion rate and geometric mean folds increase in HAI titer. | Immunogenicity profile was assessed before vaccination, 4 weeks after the vaccination and at the end of gestation period. Moreover, the HAI titer of the cord blood was also measured and compared with the maternal blood sample.
  The primary endpoint will be the seroprotection rate which is defined as the proportion of subjects with HAI titer ≥ 1:40. The other immunogenicity endpoints include seroconversion rate and geometric mean folds increase in HAI titer. Immunogenicity profile will be assessed before vaccination, 4 weeks after the vaccination and at the end of gestation period.

SECONDARY OUTCOMES:
The secondary endpoint is to evaluate the safety and tolerability profiles including the presence or absence of the pre-specified reactogenicity events and other serious/non-serious adverse events of the AdimFlu-S. | The safety information is collected from the day of vaccination to 8 weeks after the delivery.
  Safety outcomes include immediate reactions at the time of vaccination, solicited local and systemic reactions for 7 days, unsolicited adverse events until the first post-vaccination serum collected (Day 28), and serious adverse events and adverse events of special interest until 8 weeks after the delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lin SY, Wu ET, Lin CH, Shyu MK, Lee CN. The safety and immunogenicity of trivalent inactivated influenza vaccination: a study of maternal-cord blood pairs in Taiwan. PLoS One. 2013 Jun 6;8(6):e62983. doi: 10.1371/journal.pone.0062983. Print 2013. PMID 23762229